CLINICAL TRIAL: NCT01340846
Title: A Four-Part, Open-Label Study to Evaluate the Effects of Repeat Dose GSK2118436 on the Single Dose Pharmacokinetics of Warfarin, the Effects of Repeat Dose Oral Ketoconazole and Oral Gemfibrozil on the Repeat Dose Pharmacokinetics of GSK2118436, and the Repeat Dose Pharmacokinetics of GSK2118436 in Subjects With BRAF Mutant Solid Tumors
Brief Title: A Pharmacokinetics Study of the Effects of GSK2118436 on Warfarin, the Effects of Ketoconazole and Gemfibrozil on GSK2118436, and the Effects of Repeat Doses of GSK2118436 in Subjects With BRAF Mutant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113771
Record Dates: First submitted 2011-04-14; First posted 2011-04-25 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: gemfibrozil; BRAF; Drug Interactions; GSK2118436; warfarin; ketoconazole; BRAF inhibitor; oncology; BRAF positive tumor
MeSH Terms: conditions — Neoplasms | interventions — Warfarin; Ketoconazole; Gemfibrozil; dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A (Experimental): Warfarin dosed at 15mg
  Interventions: Drug: Warfarin; Drug: GSK2118436 150mg
- Part B (Experimental): Ketoconazole dosed at 400mg
  Interventions: Drug: Ketoconazole; Drug: GSK2118436 75mg
- Part C (Experimental): Gemfibrozil dosed at 600mg
  Interventions: Drug: Gemfibrozil; Drug: GSK2118436 75mg
- Part D (Experimental): GSK2118436 dosed alone
  Interventions: Drug: GSK2118436 150mg

INTERVENTIONS:
Drug: Warfarin — Warfarin dosed at 15mg on Day 1 and Day 22
  Arms: Part A
Drug: Ketoconazole — Ketoconazole dosed at 400mg daily on Days 19 through 22
  Arms: Part B
Drug: Gemfibrozil — Gemfibrozil dosed at 600mg twice daily on Days 19 through 22
  Arms: Part C
Drug: GSK2118436 150mg — GSK2118436 dosed at 150mg twice daily
  Arms: Part A; Part D
Drug: GSK2118436 75mg — GSK2118436 dosed at 75mg twice daily
  Arms: Part B; Part C

SUMMARY:
GSK2118436 is an orally administered, potent and selective small molecule BRAF inhibitor that is being developed for the treatment of BRAF mutation-positive tumors. This is a 4-part study (in 4 separate cohorts of subjects) designed to examine the interaction potential of GSK2118436, either as a perpetrator (i.e., effect of GSK2118436 on warfarin; Part A) or victim (i.e., effect of other drugs on GSK2118436; Part B: ketoconazole and Part C: gemfibrozil), as well as to evaluate the single and repeat dose pharmacokinetic parameters of GSK2118436 (Part D). A sufficient number of subjects will be screened to obtain approximately 12 evaluable subjects each for Part A, Part B, Part C and Part D. Following completion of this study, subjects may continue dosing with GSK2118436 in the roll-over study, Protocol BRF114144.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age at the time of signing the informed consent form;
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form;
* Body weight >/= 45 kg and a body mass index >/= 19 kg/m2 and </= 35 kg/m2 (inclusive);
* Able to swallow and retain oral medication;
* BRAF V600 mutation-positive tumor as determined in a CLIA-approved laboratory or equivalent (the local BRAF testing may be subject to subsequent verification by centralized testing);
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1; NOTE: Subjects with a performance status of 2 can be enrolled if the patient's confinement to bed and inability to carry out work activities is due solely to cancer-related pain, as assessed by the Investigator;
* Women of child-bearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control. Additionally, women of childbearing potential must have a negative serum pregnancy test within 14 days prior to the first dose of study medication;
* Must have adequate organ function as defined by the following values:

Absolute neutrophil count (ANC) >/=1.2 x 109/L Hemoglobin >/= 9 g/dL Platelets >/= 100 x 109/L Serum bilirubin >/= 1.5 x Upper Limit of Normal (ULN) AST and ALT >/= 2.5 x ULN; <5 x ULN if liver metastases are present (with approval of GSK medical monitor) Serum creatinine >/= ULN or calculated creatinine clearance >/= 60 mL/min PT/INR and partial thromboplastin time (PTT) >/= 1.3 x ULN Left ventricular ejection fraction >/= institutional lower limit of normal by ECHO

* CYP2C9 genotype of *1/*1 (wildtype), *1/*2 or *1/*3 (Part A only)

Exclusion Criteria:

* Currently receiving cancer therapy (e.g., chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy) within the last three weeks; chemotherapy regimens without delayed toxicity within the last 2 weeks;
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 28 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is warranted by the data);
* Current use of a prohibited medication or herbal preparation or requires any of these medications during the study;
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication;
* History of sensitivity to heparin or heparin-induced thrombocytopenia;
* Any major surgery within the last 4 weeks;
* Unresolved toxicity greater than National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI CTCAE v4.0) [NCI, 2009] Grade 2 from previous anti-cancer therapy except alopecia;
* Presence of active GI disease or other condition (e.g., small bowel or large bowel resection) that will interfere significantly with the absorption of drugs. If clarification is needed as to whether a condition will significantly affect absorption of drugs, contact the GSK medical monitor;
* A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence of HBV clearance may be enrolled);
* Presence of invasive malignancy, other than the primary diagnosis;
* Parts B and C: Subjects with brain metastases are excluded if their brain metastases are either:

Symptomatic Treated (surgery, radiation therapy) but not clinically and radiographically stable one month after local therapy, or Asymptomatic and untreated but > 1 cm in the longest dimension Patients with small (≤ 1 cm in the longest dimension), asymptomatic brain metastases that do not need immediate local therapy can be enrolled with the approval of the GSK medical monitor. Subjects on a stable dose of corticosteroids for more than one month, or those who have been off corticosteroids for at least two weeks can be enrolled. Subjects must also be off of enzyme-inducing anticonvulsants for more than four weeks; Note: Any brain metastases is exclusionary for Part A (must be excluded by prior imaging);

* Corrected QT (QTcB) interval >/= 480 msecs;
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 24 weeks;
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; abnormal cardiac valve morphology documented by ECHO (subjects with minimal abnormalities [i.e., mild regurgitation/stenosis] can be entered on study - if clarification is needed as to whether an ECHO abnormality is minimal, please contact the GSK medical monitor); or history of known cardiac arrhythmias (except sinus arrythmias) within the past 24 weeks;
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drugs, or excipients (note: to date there are no known drugs chemically related to GSK2118436 which are approved by the FDA);
* Uncontrolled medical conditions (e.g., diabetes mellitus, hypertension, liver disease), psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol;
* Subjects with known glucose 6 phosphate dehydrogenase (G6PD) deficiency;
* Pregnant females as determined by positive hCG test at screening or prior to dosing;
* Lactating females who are actively breast feeding;
* Subject is mentally or legally incapacitated;
* Part A only: Use of warfarin or exogenous Vitamin K (other than from dietary sources) within 30 days prior to treatment with study medication;
* Part A only: Subjects with history of GI bleeding, or GI ulceration;
* Part A only: Subjects with known history of Protein C and/or Protein S deficiency, or any other type of coagulopathy;
* Part A only: Subjects requiring any type of anticoagulation, or taking Aspirin at doses greater than 81 mg/day;
* Part A only: Subjects with brain metastases;
* Part A only: Any subject who by history regularly consumes a large quantity of foods rich in vitamin K will be excluded unless he/she restricts the vitamin K intake for at least one week prior to the first dose of warfarin. For study purposes, large quantities of vitamin K-containing food will be defined as 10 or more portions per week of the following: kale, spinach, turnip greens, cauliflower, chick peas, brussels sprouts, green tea, liver, soybean oil and soy protein products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-09-03 (Actual); Primary Completion 2012-11-14 (Actual); Study Completion 2012-11-14 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of S-warfarin with and without GSK2118436 | Up to 168 hours after dosing on Day 1 (warfarin alone) and Day 22 (warfarin in combination with GSK2118436)
Area under the concentration time curve (AUC) of S-warfarin with and without GSK2118436 | Up to 168 hours after dosing on Day 1 (warfarin alone) and Day 22 (warfarin in combination with GSK2118436)
Maximum plasma concentration (Cmax) of GSK2118436 with and without an inhibitor | Up to 12 hours after dosing on Day 18 (GSK2118436 alone) and Day 22 (GSK2118436 in combination with inhibitor)
Area under the concentration time curve (AUC) of GSK2118436 with and without an inhibitor | Up to12 hours after dosing on Day 18 (GSK2118436 alone) and Day 22 (GSK2118436 in combination with inhibitor)
Cmax of GSK2118436 and metabolites after single and multiple 75mg HPMC dose | Up to 24 hours after dosing on Day 1 and up to 12 hours after dosing on Day 18
AUC of GSK2118436 and metabolites after single and multiple 75mg HPMC dose | Up to 24 hours after dosing on Day 1 and up to 12 hours after dosing on Day 18
Time to Cmax (Tmax) of GSK2118436 and metabolites after single and multiple 75mg HPMC dose | Up to 24 hours after dosing on Day 1 and up to 12 hours after dosing on Day 18
Half-life of GSK2118436 and metabolites after single 75mg HPMC dose | Up to 24 hours after dosing on Day 1
Cmax of GSK2118436 and metabolites after single and multiple 150mg HPMC dose | Up to 24 hours after dosing on Day 1 and up to 12 hours after dosing on Day 18
AUC of GSK2118436 and metabolites after single and multiple 150mg HPMC dose | Up to 24 hours after dosing on Day 1 and up to 12 hours after dosing on Day 18
Tmax of GSK2118436 and metabolites after single and multiple 150mg HPMC dose | Up to 24 hours after dosing on Day 1 and up to 12 hours after dosing on Day 18
Half-life of GSK2118436 and metabolites after single 150mg HPMC dose | Up to 24 hours after dosing on Day 1

SECONDARY OUTCOMES:
Cmax of R-warfarin with and without GSK2118436 | Up to 168 hours after dosing on Day 1 (warfarin alone) and Day 22 (warfarin in combination with GSK2118436)
Time to Cmax (Tmax) of R-warfarin | Up to 168 hours after dosing on Day 1 (warfarin alone) and Day 22 (warfarin in combination with GSK2118436)
Trough concentration of GSK2118436 | Up to168 hours after dosing on Day 22
Number of subjects with adverse events as a measure of safety and tolerability | From date of first dose to transition to Rollover protocol BRF114144 (22 - 29 days) or study follow up visit if subject does not transition to BRF114144 (approximately 29 - 39 days)
Tmax for GSK2118436 with and without an inhibitor | Up to 12 hours after dosing on Day 18 (GSK2118436 alone) and Day 22 (GSK2118436 in combination with inhibitor)
AUC, Cmax, Tmax and trough concentration of GSK2118436 metabolites with and without an inhibitor, and AUC ratio of metabolites to parent | Up to 12 hours after dosing on Day 18 (GSK2118436 alone) and Day 22 (GSK2118436 in combination with inhibitor)
Inhibitor concentrations in combination with GSK2118436 | Up to12 hours after dosing on Day 22 (GSK2118436 in combination with inhibitor)
AUC of R-warfarin with and without GSK2118436 | Up to 168 hours after dosing on Day 1 (warfarin alone) and Day 22 (warfarin in combination with GSK2118436)
Terminal half-life (t1/2) of R-warfarin | Up to 168 hours after dosing on Day 1 (warfarin alone) and Day 22 (warfarin in combination with GSK2118436)
Cmax of GSK2118436 | Up to168 hours after dosing on Day 22
Trough concentration for GSK2118436 with and without an inhibitor | Up to 12 hours after dosing on Day 18 (GSK2118436 alone) and Day 22 (GSK2118436 in combination with inhibitor)
Cmax of GSK2118436 metabolites with and without an inhibitor | Up to 12 hours after dosing on Day 18 (GSK2118436 alone) and Day 22 (GSK2118436 in combination with inhibitor)
Tmax of GSK2118436 metabolites with and without an inhibitor | Up to 12 hours after dosing on Day 18 (GSK2118436 alone) and Day 22 (GSK2118436 in combination with inhibitor)
Trough concentration of GSK2118436 metabolites with and without an inhibitor | Up to 12 hours after dosing on Day 18 (GSK2118436 alone) and Day 22 (GSK2118436 in combination with inhibitor)
AUC ratio of metabolites to parent with and without an inhibitor | Up to 12 hours after dosing on Day 18 (GSK2118436 alone) and Day 22 (GSK2118436 in combination with inhibitor)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (8):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Salt Lake City, Utah
- GSK Investigational Site, Nedlands, Western Australia, Australia
- United Kingdom (2):
  - GSK Investigational Site, Headington
  - GSK Investigational Site, London

REFERENCES:
- See also: Results for study 113771 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113771?search=study&study_ids=113771#rs